CLINICAL TRIAL: NCT02142686
Title: Comparison Between Different Filling Pressures in Diagnostic Outpatient Hysteroscopy: A Double Blinded Randomised Controlled Trial.
Brief Title: Comparison Between Different Filling Pressures in Diagnostic Outpatient Hysteroscopy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, AbdelGany Hassan, Lecturer, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Supportive Care
Other Study IDs: Hyst 1
Record Dates: First submitted 2014-05-16; First posted 2014-05-20 (Estimated); Last update posted 2016-01-27 (Estimated); Status verified 2016-01

CONDITIONS: Hysteroscopy
Keywords: Hysteroscopy; Filling pressures

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Filling pressure 80 (Active Comparator): After the hysteroscope is introduced into the uterine cavity, the filling pressure will remain at 80mm.
  Interventions: Device: Filling pressure 80
- Filling pressure 50. (Active Comparator): After the hysteroscope is introduced into the uterine cavity, the filling pressure will be reduced to 50mm Hg in this group
  Interventions: Device: Filling pressure 50
- illing pressure 30 (Active Comparator): After the hysteroscope is introduced into the uterine cavity, the filling pressure will be reduced to 30mm Hg.
  Interventions: Device: Filling pressure 30

INTERVENTIONS:
Device: Filling pressure 80 — After the hysteroscope is introduced into the uterine cavity, the filling pressure will remain at 80mm Hg.
  Arms: Filling pressure 80
Device: Filling pressure 50 — After the hysteroscope is introduced into the uterine cavity, the filling pressure will be reduced to 50mm Hg.
  Arms: Filling pressure 50.
Device: Filling pressure 30 — After the hysteroscope is introduced into the uterine cavity, the filling pressure will be reduced to 30mm
  Arms: illing pressure 30

SUMMARY:
The aim of this study is to compare different filling pressures

DETAILED DESCRIPTION:
This study is a prospective double blinded randomised controlled trial. 240 women will be randomly divided into 3 groups, each containing 70 women. Randomisation will be performed using a computer generated random numbers and sealed envelopes.

Full history will be taken followed by general and local examination. The procedure will be done in the lithotomy position. Hysteroscopy will be done using a 5mm outer diameter continuous flow hysteroscope with a French working channel and a 30 degrees direction of view provided by Techno GmbH and CO. The hysteroscope will be introduced using the vaginoscopy technique, in which no speculum will be used. The cervix will be detected and the external os will be identified using the hysteroscope. The hysteroscope will be introduced in the uterine cavity. Saline will be used as the distension medium and the pressure will be set at 80mm Hg until the hysteroscope is introduced in the uterine cavity. After the hysteroscope is introduced into the uterine cavity, the filling pressure will remain at 80mm Hg in group1, will be reduced to 50mm Hg in group 2 and to 30mmHg in group 3. Randomisation will be double blind; neither the operator nor the patient will know the pressure during the procedure, a third party will set the pressure according to the computer generated random numbers.

The anterior wall, posterior wall and tubal ostea will be visualised, any polyps, adhesions septa, congenital malformations or submucous fibroids will be noted.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-60 years
* Has a clear Indication to have an outpatient hysteroscopy
* Consent to participate in the study

Exclusion Criteria:

* Premenstrual and midmenstrual patients.
* Patients with missed periods.
* Patients with known cardiac disease.
* Patients who need operative hysteroscopy

Ages: 18 Years to 60 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 240 (Actual)
Dates: Start 2014-05; Primary Completion 2015-04 (Actual); Study Completion 2015-04 (Actual)

PRIMARY OUTCOMES:
adequate visualization of the uterine cavity | 10 minutes after starting the procedure.
  10 minutes after starting the procedure, the operator will document if adequate visualization was achieved using the allocated pressure. If visualization was not adequate, he will document that adequate visualization was not achieved using the allocated pressure and will ask for the pressure to be adjusted.

SECONDARY OUTCOMES:
Pain perceived by the patient | 10 minutes after starting the procedure
  Pain will be assessed by a visual analogue scale 10 minutes after starting the procedure.
Pain perceived by the patient 30 minutes after starting the procedure. | 30 minutes after starting the procedure.
  Pain will be assessed by a visual analogue scale 30 minutes after starting the procedure.

CONTACTS AND LOCATIONS:
Overall Officials: AbdelGany M A Hassan, MRCOG, MD, Principal Investigator — Cairo University
Locations (1):
- Cairo University Hospitals, Cairo, Egypt

REFERENCES:
- [Background] Sharma JB, Aruna J, Kumar P, Roy KK, Malhotra N, Kumar S. Comparison of efficacy of oral drotaverine plus mefenamic acid with paracervical block and with intravenous sedation for pain relief during hysteroscopy and endometrial biopsy. Indian J Med Sci. 2009 Jun;63(6):244-52. PMID 19602758
- [Background] van Dongen H, de Kroon CD, Jacobi CE, Trimbos JB, Jansen FW. Diagnostic hysteroscopy in abnormal uterine bleeding: a systematic review and meta-analysis. BJOG. 2007 Jun;114(6):664-75. doi: 10.1111/j.1471-0528.2007.01326.x. PMID 17516956
- [Background] O'Flynn H, Murphy LL, Ahmad G, Watson AJ. Pain relief in outpatient hysteroscopy: a survey of current UK clinical practice. Eur J Obstet Gynecol Reprod Biol. 2011 Jan;154(1):9-15. doi: 10.1016/j.ejogrb.2010.08.015. PMID 20926175
- [Background] Shahid A, Pathak M, Gulumser C, Parker S, Palmer E, Saridogan E. Optimum uterine filling pressure for outpatient diagnostic hysteroscopy: a double-blind, randomized controlled trial. Reprod Biomed Online. 2014 Jan;28(1):86-91. doi: 10.1016/j.rbmo.2013.07.018. Epub 2013 Sep 14. PMID 24262433